CLINICAL TRIAL: NCT07275853
Title: A Phase I Clinical Study of KXV01 TCR Lentinvivo Injection on Safety, Tolerability, and Efficacy in Patients With Advanced Solid Tumors
Brief Title: Personalized KXV01 Lentinvivo (TCR) Injection as the Therapy for Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TCRx Therapeutics Co.Ltd (Industry)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KXV01-R101-08
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KXV01 TCR Lentinvivo Injection (Experimental): KXV01 TCR Lentinvivo Injection
  Interventions: Drug: KXV01 TCR Lentinvivo Injection

INTERVENTIONS:
Drug: KXV01 TCR Lentinvivo Injection — KXV01 TCR Lentinvivo Injection is one kind of third-generation non-replicative self-inactivating lentivirus vector which carries an effective patient's personalized tumor-reactive TCR.

SUMMARY:
This is a single center, single arm, open-label, dose escalation, phase 1 study to evaluate the safety, tolerability and preliminary efficacy of KXV01 TCR Lentinvivo for patients with advanced solid tumors.

DETAILED DESCRIPTION:
In recent years, the field has found that patient-specific anti-tumor treatment technologies have increasingly significant clinical application prospects and clinical value. Patient-specific anti-tumor in vivo TCR gene therapy is an advanced therapeutic strategy that can specifically recognize tumor neoantigens. This strategy is not restricted by patients' HLA typing nor by the type of indication.

This investigator-initiated clinical study aims to evaluate KXV01 TCR Lentinvivo, the third-generation self-inactivating lentiviral vector that carries patient-derived personalized tumor reactive TCR, in patients with advanced solid tumors. The study employs a BOIN design to assess safety, tolerability, and preliminary efficacy.

ELIGIBILITY:
Screening Period 1

Inclusion Criteria 1:

1. Voluntarily participate in the clinical study; fully understand the study and voluntarily sign the informed consent form; be willing to comply with and able to complete all trial procedures.
2. Aged 18 to 70 years (inclusive).
3. Histologically or cytologically confirmed incurable or metastatic solid tumors that have failed standard treatment, or for which no standard treatment is currently available.
4. Expected survival time > 6 months.
5. ECOG performance status of 0 or 1.
6. Sufficient organ function, defined as follows:

   6.1) Hematological system: 6.1.1) Hemoglobin ≥ 90 g/L (no blood transfusion within 14 days prior to the test); 6.1.2) Absolute neutrophil count ≥ 1.5 × 10⁹/L (no granulocyte colony-stimulating factor treatment within 14 days prior to the test); 6.1.3) Platelet count ≥ 100 × 10⁹/L in the absence of significant hepatic lesions (primary or metastatic) (no platelet transfusion within 14 days prior to the test), or ≥ 75 × 10⁹/L in the presence of hepatic lesions (no platelet transfusion within 14 days prior to the test); 6.1.4) Absolute lymphocyte count (ALC) ≥ 0.7 × 10⁹/L; 6.2) Hepatic function: 6.2.1) Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN) in the absence of significant hepatic lesions (primary or metastatic), and ≤ 3 × ULN in subjects with hepatic lesions or Gilbert's disease; 6.2.2) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN (≤ 5 × ULN in subjects with liver metastasis or liver cancer); alkaline phosphatase (ALP) ≤ 2.5 × ULN (≤ 5 × ULN in subjects with bone metastasis); 6.3) Renal function: Creatinine clearance ≥ 60 mL/min (Cockcroft-Gault formula: ([140 - age] × weight [kg] × [0.85, for females only]) / (72 × creatinine (mg/dl))); 6.4) Baseline oxygen saturation > 92% during natural breathing (without auxiliary oxygen supply).
7. Patients whose tumor lesions can be collected and from whom tumor-reactive TCR sequences can be identified may enter the study. If a patient has obtained individualized TCR sequences from previously collected archived tumor tissue in other studies, they may directly enter Screening Period 2, provided that the archived tissue was collected within one year prior to signing the informed consent form for this study.
8. Women of childbearing age must have a negative urine/blood pregnancy test during the screening period and agree to use contraceptive measures for at least 1 year after administration; male subjects whose partners are of childbearing potential must agree to use effective barrier contraception for at least 1 year after administration.

Exclusion Criteria 1:

1. A history of other malignant tumors within 2 years prior to signing the informed consent form, except for non-melanoma skin cancer, some in situ carcinomas (e.g., cervical cancer, bladder cancer, breast cancer), or low-risk prostate cancer.
2. Uncontrolled infectious diseases within 4 weeks prior to signing the informed consent form.
3. Active hepatitis B or hepatitis C virus infection.
4. Patients with HIV infection.
5. Patients with positive Treponema pallidum.
6. A history of any of the following cardiovascular diseases within the past 6 months: New York Heart Association (NYHA) Class III or IV heart failure, coronary angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant heart diseases.
7. Tumor lesions invading the heart or major blood vessels.
8. Abnormal pulmonary function indicated by a ratio of forced expiratory volume in 1 second (FEV1) to forced vital capacity (FVC) < 70% in pulmonary function tests.
9. A history of clinically significant central nervous system (CNS) disorders, including but not limited to epilepsy, paresis, aphasia, stroke, severe traumatic brain injury, dementia, Parkinson's disease, cerebellar disease, and organic brain syndrome.
10. Use of the following drugs or treatments:

    1. Hormones: Use of therapeutic doses of corticosteroids (defined as prednisone or equivalent > 20 mg/day) within 72 hours prior to administration of the study drug; physiologic replacement doses, topical, and inhaled steroids are permitted;
    2. Chemotherapy: Receipt of salvage chemotherapy within 2 weeks prior to administration of the study drug;
    3. GvHD treatment: Receipt of anti-GvHD therapy within 4 weeks prior to administration of the study drug;
    4. Allogeneic bone marrow transplantation;
    5. Gene therapy;
    6. Adoptive cell therapy;
11. Females who are pregnant or breastfeeding.
12. A history of primary immunodeficiency or autoimmune disease, except for the following:

    * History of hypothyroidism with stable thyroid hormone replacement therapy;
    * Patients with well-controlled type 1 diabetes mellitus.
13. Patients whose disease or condition renders them unable to understand, participate in, and/or comply with the study protocol.
14. Any other disease that the investigator believes would impair the subject's ability to tolerate protocol treatment or significantly increase the risk of complications.
15. Current or past history of psychoactive substance abuse or dependence.
16. Subjects whose underlying condition, in the investigator's judgment, may increase the risk of receiving the investigational drug or confound the interpretation of toxic reactions and adverse events.
17. Other conditions deemed unsuitable for participation in the study by the investigator.

Screening Period 2

Inclusion Criteria 2:

The patient's organ function and key test items at this stage should not have significant changes compared with their test results in Screening Period 1. If the patient's test results in Screening Period 2 exceed the following criteria, they should not receive administration of KXV01 Injection until the abnormal items return to the normal range.

1. The patient's KXV01 Injection has been successfully prepared.
2. Expected survival time > 6 months.
3. ECOG performance status of 0 or 1.
4. Sufficient organ function.
5. Females of childbearing potential have a negative blood pregnancy test within 7 days prior to administration of the study drug (Non-childbearing potential: surgically sterilized or postmenopausal for at least 2 years). In addition, female subjects of childbearing potential must use medically approved contraceptive measures for 12 months after the start of study treatment and have no egg retrieval during this period.
6. Male subjects are willing to use medically approved contraceptive measures from the time of signing the informed consent form until 12 months after the start of study treatment, and will not donate sperm during this period.
7. At least one measurable lesion according to RECIST v1.1 criteria.
8. Toxicities and adverse reactions caused by prior therapy should have resolved to Grade ≤ 1 (except for toxicities considered clinically insignificant, such as chemotherapy-induced alopecia).

Exclusion Criteria 2:

1. Prior to administration of the study drug, the subject's anti-tumor therapy has not been sufficiently washed out (2 weeks or 5 half-lives, whichever is shorter):

   Except for the following:
   * Gonadotropin (GnRH) agonists or antagonists used for the treatment of prostate cancer
   * Hormone replacement therapy, or oral contraceptives.
2. Uncontrolled infectious diseases within the previous 4 weeks.
3. Active hepatitis B or hepatitis C virus infection.
4. Patients with HIV infection.
5. Patients with positive Treponema pallidum.
6. Tumor lesions invading the heart or major blood vessels.
7. A history of clinically significant central nervous system (CNS) disorders, including but not limited to epilepsy, paresis, aphasia, stroke, severe traumatic brain injury, dementia, Parkinson's disease, cerebellar disease, and organic brain syndrome.
8. Known primary central nervous system (CNS) malignancy or symptomatic CNS metastases.
9. Use of the following drugs or treatments between Screening Period 1 and Screening Period 2:

   1. Hormones: Use of therapeutic doses of corticosteroids (defined as prednisone or equivalent > 20 mg/day) within 72 hours prior to administration of the study drug; physiologic replacement doses, topical, and inhaled steroids are permitted;
   2. Chemotherapy: Receipt of salvage chemotherapy within 2 weeks prior to administration of the study drug;
   3. GvHD treatment: Receipt of anti-GvHD therapy within 4 weeks prior to administration of the study drug;
   4. Allogeneic bone marrow transplantation;
   5. Gene therapy;
   6. Adoptive cell therapy;
   7. Use of alemtuzumab within 6 months prior to administration of the study drug, or clofarabine or cladribine within 3 months prior to administration;
   8. Receipt of radiotherapy between Screening Period 1 and Screening Period 2. Patients are eligible only if lesions within the radiation field show progressive disease (PD), or there are measurable lesions outside the radiation field meeting RECIST v1.1 criteria on imaging assessment; if there are measurable lesions outside the radiation field, radiotherapy to other lesions must be at least 2 weeks apart from the administration date of the study drug.
10. Females who are pregnant or breastfeeding.
11. Subjects whose underlying condition, in the investigator's judgment, may increase the risk of receiving the investigational drug or confound the interpretation of toxic reactions and adverse events.
12. Receipt of major surgery (excluding diagnostic surgery) between Screening Period 1 and Screening Period 2, or expected to undergo major surgery during the study period. Subjects with planned or ongoing minor surgical procedures (such as venous access placement, etc.) are eligible for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity | 28 days after administraiton
  DLT evaluation period: The DLT evaluation period is defined as within 28 days (inclusive) after the subjects' first infusion of KXV01 injection during the dose escalation stage. All adverse events should be graded and evaluated in accordance with CTCAE v5.0. Among them, cytokine release syndrome (CRS) and immune effector cell-related neurotoxicity syndrome (ICANS) should be determined and graded in accordance with the standards of the American Society for Transplantation and Cell Therapy (ASTCT).

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No